CLINICAL TRIAL: NCT02242357
Title: Post-Marketing Surveillance Study Micardis® Plus
Brief Title: Study to Evaluate Efficacy and Tolerability of Micardis®/Micardis® Plus in Patients With Hypertension
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.427
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with hypertension
  Interventions: Drug: Micardis®; Drug: Micardis® Plus

INTERVENTIONS:
Drug: Micardis®
Drug: Micardis® Plus

SUMMARY:
Study to evaluate efficacy and tolerability of Micardis®/Micardis® Plus under usual daily-practice prescribing conditions in hypertensive patients

ELIGIBILITY:
Inclusion Criteria:

* Males and females for whom a medical antihypertensive therapy is indicated
* Age >= 18 years

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with hypertension
Sampling Method: Non-Probability Sample
Enrollment: 14553 (Actual)
Dates: Start 2003-01; Primary Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Change in morning blood pressure (office and self-measured) | up to 6 weeks

SECONDARY OUTCOMES:
Change in heart rate | up to 6 weeks
Number of patients with adverse drug reactions | up to 6 weeks
Assessment of efficacy by investigator on a 5-point scale | at week 6
Assessment of tolerability by investigator on 5-point scale | at week 6
Change in rate of morning complaints | up to 6 weeks